CLINICAL TRIAL: NCT07268001
Title: Effects of Continuous Theta Burst Stimulation to the Dorsolateral Prefrontal Cortex in Attention to Emotional Stimuli
Brief Title: Effects of Continuous Theta Burst Stimulation on Emotional Attention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cyprus (Other)
Responsible Party: Principal Investigator, Kostas Fanti, Prof. Dr., University of Cyprus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ΕΕΒΚ/ΕΠ/2019/67
Record Dates: First submitted 2025-11-24; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- cTBS over the left DLPFC (Experimental): Participants receive 1 session of continuous theta burst stimulation (cTBS) over the left dorsolateral prefrontal cortex (DLPFC; F3, following standard coordinates from the EEG International 10-20 system). The TBS sesssion consisted of 3 pulses at 50 Hz, with each train being repeated every 200 ms (5 Hz) for 40 seconds (600 pulses). After stimulation, attentional responses to pleasant and distressing images are assessed using the dot-probe task, which measures attentional bias toward emotional stimuli by presenting pairs of pleasant-neutral, distressing-neutral and neutral-neutral images. After each image pair, a dot appears in the location of one image, and participants must quickly indicate its position.
  Interventions: Device: Continuous theta burst stimulation
- cTBS over the right DLPFC (Experimental): Participants receive 1 session of continuous theta burst stimulation (cTBS) over the right dorsolateral prefrontal cortex (DLPFC; F4, following standard coordinates from the EEG International 10-20 system). The TBS sesssion consisted of 3 pulses at 50 Hz, with each train being repeated every 200 ms (5 Hz) for 40 seconds (600 pulses). After stimulation, attentional responses to pleasant and distressing images are assessed using the dot-probe task, which measures attentional bias toward emotional stimuli by presenting pairs of pleasant-neutral, distressing-neutral and neutral-neutral images. After each image pair, a dot appears in the location of one image, and participants must quickly indicate its position.
  Interventions: Device: Continuous theta burst stimulation
- sham cTBS over the left DLPFC (Sham Comparator): Participants receive 1 session of sham continuous theta burst stimulation (cTBS) over the left dorsolateral prefrontal cortex (DLPFC; F3, following standard coordinates from the EEG International 10-20 system). Sham stimulation was delivered using a sham coil that produced the same stimulation noise, but inducing nearly zero electric-field under the coil's center. After sham stimulation, attentional responses to pleasant and distressing images are assessed using the dot-probe task, which measures attentional bias toward emotional stimuli by presenting pairs of pleasant-neutral, distressing-neutral and neutral-neutral images. After each image pair, a dot appears in the location of one image, and participants must quickly indicate its position.
  Interventions: Device: Sham Control
- sham cTBS over the right DLPFC (Sham Comparator): Participants receive 1 session of sham continuous theta burst stimulation (cTBS) over the right dorsolateral prefrontal cortex (DLPFC; F3, following standard coordinates from the EEG International 10-20 system). Sham stimulation was delivered using a sham coil that produced the same stimulation noise, but inducing nearly zero electric-field under the coil's center. After sham stimulation, attentional responses to pleasant and distressing images are assessed using the dot-probe task, which measures attentional bias toward emotional stimuli by presenting pairs of pleasant-neutral, distressing-neutral and neutral-neutral images. After each image pair, a dot appears in the location of one image, and participants must quickly indicate its position.
  Interventions: Device: Sham Control

INTERVENTIONS:
Device: Continuous theta burst stimulation — A TBS session burst consist of 3 pulses at 50 Hz, with each train being repeated every 200 ms (5 Hz) for 40 seconds (600 pulses).
  Other Names: Non invasive brain stimulation
  Arms: cTBS over the left DLPFC; cTBS over the right DLPFC
Device: Sham Control — Sham stimulation was delivered using an identical with the real Magstim figure of eight focal sham coil (70 mm diameter) that produced the same stimulation noise. Sham Magstim figure-of-eight coil have been found to induce nearly zero electric-field under the coil's center.
  Arms: sham cTBS over the left DLPFC; sham cTBS over the right DLPFC

SUMMARY:
The goal of this clinical trial is to examine the differential effect of continuous TBS (cTBS) over the left and right dorsolateral prefrontal cortex (DLPFC) on the facilitation of attention towards emotional (i.e., pleasant and distress-ing) versus neutral stimuli in healthy young adults. The main questions it aims to answer are:

1. To what extend a temporary modulation of DLPFC activity through cTBS influences attentional responses to emotional stimuli?
2. To what extend the effects of cTBS on attentional responses to emotional stimuli differ depending on whether the left or right dorsolateral prefrontal cortex (DLPFC) is stimulated?

Researchers will compare four stimulation conditions: 1) real cTBS on the left DLPFC, 2) real cTBS on the right DLPFC, 3) sham cTBS on the left DLPFC, and 4) sham cTBS on the right DLPFC, to see if participants receiving cTBS over the DLPFC would exhibit faster reaction times to probes replacing pleasant and distressing images, relative to a sham condition.

Participants will receive a short cTBS session (40 seconds), and after that, they will be presented with an emotional dot-probe task (computerized task).

Regarding the cTBS Protocol, coil positioning will be determined using standardized coordinates from the EEG International 10-20 system, with F4 corresponding to the right DLPFC stimulation target and F3 corresponding to the left DLPFC. The location and orientation of each participant's coil placement will be indicated on a nylon cap that participants wore throughout the single stimulation session. A figure-of-eight focal coil (70 mm diameter) will be used. The coil will be held in a fixed position by a mechanical arm and oriented so that the induced electric current flowed in a posterior-anterior direction. Stimulus intensities were set at 70% of active motor threshold (AMT). Each TBS session burst consists of 3 pulses at 50 Hz, with each train being repeated every 200 ms (5 Hz) for 40 seconds (600 pulses).

Regarding the dot-probe task is a common laboratory paradigm used to index attentional bias for emotional stimuli at early stages of information processing. It provides a quick, convenient, and inexpensive index of emotional responsiveness. The emotional pictures version of the task used in the current study presents a series of picture pairs of distressing (e.g., crying child), neutral (e.g., book) and pleasant (e.g., smiling baby) emotional content using images primarily taken from the International Affective Picture System (IAPS). This task consists of 1 block of practice stimuli (12 picture pairs) followed by 3 experi-mental blocks, each containing 12 picture pairs. Each picture presentation had three sequential components: (1) a 500 millisecond image of fixation cross appearing in the center of the screen, (2) a 500 millisecond simultaneous presentation of one of three potential picture pairings: neutral-neutral, pleasant-neutral and distress-neutral, with stimuli centered and located above or below the location of the fixation cross, and (3) a second image of fixation cross appearing in either the top or bottom picture location. Participants will be instructed to respond as fast as they could and after every trial they selected a key on the keyboard that corresponded to the location on the screen (up or down) where the dot-probe appeared. If no key was pressed within 5000 milliseconds, the response will be recorded as incorrect.

ELIGIBILITY:
Inclusion Criteria:

* Medication-free, right-handed, normal vision, without ant estabished risk factor to rTMS (screening performed with Transcranial Magnetic Stimulation Safety Questionnaire).

Exclusion Criteria:

* History of psychiatric/neurological disorders, such as epilepsy, head trauma and migraine.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-05-16 (Actual); Study Completion 2020-05-16 (Actual)

PRIMARY OUTCOMES:
Response times in the dot-probe task | From enrollment to the end of dot-probe task, that was performed in 1 session (1 day).
  Response times to distressing, pleasant, and neutral stimuli were assessed using the dot-probe paradigm.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No